CLINICAL TRIAL: NCT04187027
Title: Efficacy Of Pulsed Electromagnetic Field Therapy On Neurogenic Bladder in Children With Myelomeningocele
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohammed E. Ali, Lecturer, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002423
Record Dates: First submitted 2019-11-26; First posted 2019-12-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Neurogenic Bladder
Keywords: Myelomeningocele; Pulsed electromagnetic field therapy
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Meningomyelocele

STUDY DESIGN:
Intervention Model Description: Patients were divided randomly into two groups. Group (A) which is the control group received medical care and standard urotherapy only. And Group (B) which is the study group received medical care and standard urotherapy in addition to pulsed electromagnetic field therapy for three successful months. All children were assisted using urodynamic studies before and after three months of intervention.
Who Masked: Outcomes Assessor
Masking Description: Blinding process to participants and care providers was impossible due to the nature of intervention therapy. Data were analyzed by an impartial statistician (outcomes assessor), referring to each arm with an encoded name: Group A (control group) and Group B (study group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the medical care and standard care only group (No Intervention): Group (A) received medical care and standard urotherapy only.
- the medical care and standard care + P.E.M.F group (Experimental): Group (B) which received the same medical care and standard urotherapy in addition to pulsed electromagnetic field therapy that applied for 20 min, ,three times / weak for three successful months.
  Interventions: Device: pulsed electromagnetic field therapy device

INTERVENTIONS:
Device: pulsed electromagnetic field therapy device — magnetic field stimulation (MFS) is a novel technique for stimulating the nervous system non-invasively, which can activate deep neural structures via induced electric currents, without pain and discomfort. Also, several clinical trials including placebo-controlled studies have shown that MFS of the pelvic floor and sacral roots is effective for overactive bladder (OAB). MFS induces inhibitory effects on detrusor overactivity in a similar manner to electrical stimulation, with significant clinical advantages. MFS of the sacral nerve roots could be a promising alternative treatment for OAB.
  Arms: the medical care and standard care + P.E.M.F group

SUMMARY:
This study was conducted to assess the efficacy of pulsed electromagnetic field therapy on neurogenic bladder in children with myelomeningocele .Intervention: A pretest-post test controlled study was conducted in out-patient clinic in faculty of physical therapy Cairo university.

DETAILED DESCRIPTION:
Myelomeningocele is the most common cause of neurogenic bladder in children. Bladder function in these children is affected by disordered innervation of detrusor muscle and external urethral sphincter that may lead to hydronephrosis. Thirty myelomeningocele children with neurogenic bladder were enrolled in this study and were assessed for eligibility. Their aged between 4 and 12 years. They were divided randomly into two groups. Group (A) which is the control group received medical care and standard urotherapy only. And Group (B) which is the study group received medical care and standard urotherapy in addition to pulsed electromagnetic field therapy for three successful months. All children were assisted using urodynamic studies before and after three months of intervention.

ELIGIBILITY:
Inclusion Criteria:

* their age was ranging from four to twelve years.
* children participated in this study were from both sexes.
* all children with stable medical and psychological status and had the same socioeconomic status.
* they were able to follow the verbal commands or instructions.

Exclusion Criteria:

* children with visual or auditory problems.
* children with any neurological manifestation rather than spina bifida.
* medically unstable children especially with cardiovascular disorders, or mentally retarded children.
* children with any sign of urinary tract infection, or any implanted metal.
* uncooperative children.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2025-05-27 (Actual); Primary Completion 2025-11-19 (Actual); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
The mean (SD) maximum urinary flow rate (Q max) | maximum urinary flow rate (Q max) was assessed at day 0.
  Measurement of maximum urinary flow rate (Qmax) is widely used in the assessment of men complaining of lower urinary tract symptoms (LUTS). Although Qmax varies with age and voided volume (V. void), a reduced flow rate can be used clinically to suggest the presence of bladder outlet obstruction (BOO).
The mean (SD) maximum urinary flow rate (Q max) | maximum urinary flow rate (Q max) was assessed at day 90.
  Measurement of maximum urinary flow rate (Qmax) is widely used in the assessment of men complaining of lower urinary tract symptoms (LUTS). Although Qmax varies with age and voided volume (V. void), a reduced flow rate can be used clinically to suggest the presence of bladder outlet obstruction (BOO).
The mean (SD) maximum cystometric capacity (MCC) | maximum cystometric capacity (MCC) was assessed at day 0.
  Maximum cystometric capacity in patients with normal sensation, is the volume at which the patient feels he/she can no longer delay micturition (has a strong desire to void)
The mean (SD) maximum cystometric capacity (MCC) | maximum cystometric capacity (MCC) was assessed at day 90.
  Maximum cystometric capacity in patients with normal sensation, is the volume at which the patient feels he/she can no longer delay micturition (has a strong desire to void)
The mean (SD) of incidence of first uninhibited detrusor contraction | first uninhibited detrusor contraction was assessed at day 0.
  Detrusor hyperreflexia (DH) is a frequently occurring condition. The symptomatology is characterized by frequency, urgency and urge incontinence. DH is defined as involuntary, uninhibited detrusor contractions
The mean (SD) of incidence of first uninhibited detrusor contraction | first uninhibited detrusor contraction was assessed at day 90.
  Detrusor hyperreflexia (DH) is a frequently occurring condition. The symptomatology is characterized by frequency, urgency and urge incontinence. DH is defined as involuntary, uninhibited detrusor contractions

CONTACTS AND LOCATIONS:
Overall Officials: Nehad A. Abo-zaid, PhD, Principal Investigator — South Valley University, Faculty of Physical Therapy; Mohammed E. Ali, PhD student, Principal Investigator — South Valley University, Faculty of Physical Therapy
Locations (2):
- Egypt (2):
  - South Valley University, Faculty of Physical Therapy, Qina, Qena Governorate
  - Faculty of Physical Therapy, Outpatient Clinic, Qina, Qena Governorate

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choe JH, Choo MS, Lee KS. Symptom change in women with overactive bladder after extracorporeal magnetic stimulation: a prospective trial. Int Urogynecol J Pelvic Floor Dysfunct. 2007 Aug;18(8):875-80. doi: 10.1007/s00192-006-0261-0. Epub 2006 Nov 30. PMID 17136485
- [Background] Sheriff MK, Shah PJ, Fowler C, Mundy AR, Craggs MD. Neuromodulation of detrusor hyper-reflexia by functional magnetic stimulation of the sacral roots. Br J Urol. 1996 Jul;78(1):39-46. doi: 10.1046/j.1464-410x.1996.00358.x. PMID 8795398
- [Background] Ikeda Y, Fry C, Hayashi F, Stolz D, Griffiths D, Kanai A. Role of gap junctions in spontaneous activity of the rat bladder. Am J Physiol Renal Physiol. 2007 Oct;293(4):F1018-25. doi: 10.1152/ajprenal.00183.2007. Epub 2007 Jun 20. PMID 17581924
- [Background] Dorsher PT, McIntosh PM. Neurogenic bladder. Adv Urol. 2012;2012:816274. doi: 10.1155/2012/816274. Epub 2012 Feb 8. PMID 22400020
- [Background] Fergany LA, Shaker H, Arafa M, Elbadry MS. Does sacral pulsed electromagnetic field therapy have a better effect than transcutaneous electrical nerve stimulation in patients with neurogenic overactive bladder? Arab J Urol. 2017 Mar 29;15(2):148-152. doi: 10.1016/j.aju.2017.01.007. eCollection 2017 Jun. PMID 29071144
- [Background] Madersbacher H. Neurogenic bladder dysfunction in patients with myelomeningocele. Curr Opin Urol. 2002 Nov;12(6):469-72. doi: 10.1097/00042307-200211000-00004. PMID 12409874
- [Result] Baradaran N, Ahmadi H, Nejat F, El Khashab M, Mahdavi A. Nonneural congenital abnormalities concurring with myelomeningocele: report of 17 cases and review of current theories. Pediatr Neurosurg. 2008;44(5):353-9. doi: 10.1159/000149900. Epub 2008 Aug 15. PMID 18703879
- [Result] Larijani FJ, Moghtaderi M, Hajizadeh N, Assadi F. Preventing kidney injury in children with neurogenic bladder dysfunction. Int J Prev Med. 2013 Dec;4(12):1359-64. PMID 24498490
- [Result] Wu HY, Baskin LS, Kogan BA. Neurogenic bladder dysfunction due to myelomeningocele: neonatal versus childhood treatment. J Urol. 1997 Jun;157(6):2295-7. PMID 9146656
- [Result] Kim JW, Kim MJ, Noh JY, Lee HY, Han SW. Extracorporeal pelvic floor magnetic stimulation in children with voiding dysfunction. BJU Int. 2005 Jun;95(9):1310-3. doi: 10.1111/j.1464-410X.2005.05524.x. PMID 15892823
- [Result] Bycroft JA, Craggs MD, Sheriff M, Knight S, Shah PJ. Does magnetic stimulation of sacral nerve roots cause contraction or suppression of the bladder? Neurourol Urodyn. 2004;23(3):241-5. doi: 10.1002/nau.20009. PMID 15098220
- [Result] Juszczak K, Kaszuba-Zwoinska J, Thor PJ. Pulsating electromagnetic field stimulation of urothelial cells induces apoptosis and diminishes necrosis: new insight to magnetic therapy in urology. J Physiol Pharmacol. 2012 Aug;63(4):397-401. PMID 23070089
- [Result] Ellsworth P, Cone EB. Neurogenic detrusor overactivity: an update on management options. R I Med J (2013). 2013 Apr 1;96(4):38-40. PMID 23641451
- [Result] Amarante MA, Shrensel JA, Tomei KL, Carmel PW, Gandhi CD. Management of urological dysfunction in pediatric patients with spinal dysraphism: review of the literature. Neurosurg Focus. 2012 Oct;33(4):E4. doi: 10.3171/2012.7.FOCUS12232. PMID 23025445
- [Result] Quek P. A critical review on magnetic stimulation: what is its role in the management of pelvic floor disorders? Curr Opin Urol. 2005 Jul;15(4):231-5. doi: 10.1097/01.mou.0000172395.54643.4d. PMID 15928511
- [Result] Takahashi S, Kitamura T. Overactive bladder: magnetic versus electrical stimulation. Curr Opin Obstet Gynecol. 2003 Oct;15(5):429-33. doi: 10.1097/00001703-200310000-00012. PMID 14501247